CLINICAL TRIAL: NCT05499416
Title: Effect of Bimekizumab in Patients With Psoriasis Vulgaris and Active Psoriatic Arthritis Who Have an Inadequate Skin Response to Anti-IL23 Therapy
Brief Title: Effect of Bimekizumab in Patients With Psoriasis Vulgaris and Active Psoriatic Arthritis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision.
Sponsor: Innovaderm Research Inc. (Other)
Collaborators: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNO-5031
Record Dates: First submitted 2022-08-03; First posted 2022-08-12 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Psoriasis Vulgaris; Active Psoriatic Arthritis
Keywords: plaque psoriasis; systemic therapy; psoriasis vulgaris; arthritic psoriasis; bimekizumab
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bimekizumab 320 mg SC injections (Experimental): Bimekizumab 320 mg solution administered via SC injections every 4 weeks for 16 weeks.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Self-administration of two (2-160 mg/mL [1 mL]) pre-filled syringes or autoinjectors at baseline (Day1) and at Weeks 4, 8,12, and 16
  Other Names: BIMZELX®

SUMMARY:
This is an open-label study to evaluate the effects of bimekizumab in patients with psoriasis vulgaris and who also have active psoriatic arthritis (PsA).

DETAILED DESCRIPTION:
This study is being conducted to evaluate the effects of bimekizumab administered subcutaneously (SC) to patients with psoriasis vulgaris and who also have active PsA who have an inadequate skin response to anti-interleukin (IL)23 therapy. Approximately 20 adult subjects with psoriasis vulgaris and active PsA who have an inadequate skin response to anti-IL23 will receive bimekizumab 320 mg solution administered SC every 4 weeks for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient 18 years of age or older at the time of consent.
2. Patient with a history of psoriasis vulgaris and PsA (as determined by the investigator) for ≥ 6 months prior to the screening visit.
3. Patient with moderate-to-severe psoriasis vulgaris before initiating treatment with an anti-IL23 agent.
4. Patient with an inadequate skin response to at least 12 weeks treatment with an anti-IL23 agent for the treatment of psoriasis vulgaris as defined by a PGA ≥ 2 and plaque psoriasis covering ≥ 1% of total BSA (excluding palms and soles) at the screening and Day 1 visits.
5. Patient with active PsA as defined by ≥ 1 joint that is tender (TJC68) and/or swollen (SJC66) at Day 1.

Exclusion Criteria:

1. Female who is breastfeeding, pregnant, or who is planning to become pregnant during the study or within 4 months after the last study product administration.
2. Patient with evidence of erythrodermic, pustular, predominantly guttate psoriasis, or drug-induced psoriasis.
3. Patient with any known clinically significant medical condition or presence of a skin or rheumatologic disease that would, in the opinion of the investigator, put the patient at undue risk or interfere with the interpretation of study results.
4. Patient who plans to receive a live or live-attenuated vaccine during the study and up to 4 weeks or 5 half-lives (of the study product), whichever is longer, after the last study product administration.
5. Patient with an active infection (except common cold) that would place them at increased risk, a recent serious infection, or a history of opportunistic, recurrent, or chronic infections.
6. Patient with a diagnosis of inflammatory bowel disease (Crohn's disease or ulcerative colitis).
7. Patient with known or suspected hypersensitivity to bimekizumab or any component of the investigational product, including any nonmedicinal ingredient, or component of the container.
8. Patient who has received any marketed or investigational biological agent, except anti-IL23 agents, within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
9. Patient who has received treatment with bimekizumab prior to Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Physician Global Assessment (PGA) x Body Surface Area (BSA) | Week 24
  The product of physician's global assessment and body surface area (PGA×BSA) is a measure of psoriasis severity (0-400), with higher scores indicating more severe disease.
Proportion of patients achieving MDA | Week 24
  A patient will be considered to have achieved MDA when meeting 5/7 of the following criteria: tender joints count ≤ 1; swollen joints count ≤ 1; Psoriasis Area and Severity Index (PASI) ≤ 1 or body surface area (BSA) ≤ 3%; patient pain visual analog scale (VAS) ≤ 15 mm; patient's global assessment of arthritis visual analog scale (PtGA VAS) ≤ 20 mm; Health Assessment Questionnaire-Disability Index (HAQ-DI) ≤ 0.5; tender entheseal points ≤ 1.

SECONDARY OUTCOMES:
Physician Global Assessment (PGA) | Weeks 12 and 24
  The PGA is a global assessment of the current state of the disease. It is a 5-point (0-4) morphological assessment of overall disease severity, with higher scores indicating more severe disease.
Body Surface Area (BSA) | Weeks 12 and 24
  The overall BSA affected by psoriasis vulgaris will be evaluated (from 0% to 100%).
Psoriasis Area and Severity Index (PASI) | Weeks 12 and 24
  The PASI is a composite score that considers the degree of erythema, induration/infiltration, and desquamation (each scored from 0 to 4 separately) for each of 4 body regions.
American College of Rheumatology (ACR) | Week 24
  The ACR is a composite including the number of tender and number of swollen joints, patient's global assessment of arthritis visual analog scale (PtGA VAS), physician global assessment visual analog scale (MDGA VAS), Health Assessment Questionnaire-Disability Index (HAQ-DI), patient pain visual analog scale (VAS), and C-reactive protein (CRP) levels. The proportion of patients achieving ACR20, ACR50, and ACR70 will be calculated.
Tender joints count (TJC) | Week 24
  The tenderness of 68 joints (TJC68) will be assessed and the counts recorded.
Swollen joints count (SJC) | Week 24
  The level of swelling at 66 joints (SJC66) will be assessed and the counts recorded. The swollen joints count can range between 0 and 66 and represents the sum of the total number of swollen joints.
Physician's Global Assessment of Arthritis Visual Analogue Scale (MDGA VAS) | Week 24
  The physician's global assessment of disease activity will be measured using 100-mm VAS scale with anchor statements on the left (none) and on the right (extremely active).
Patient's Assessment of Arthritis Pain Visual Analogue Scale (patient pain VAS) | Week 24
  The patient's assessment of pain will be measured using 100-mm VAS scale with anchor statements on the left (no pain) and on the right.
Patient's Global Assessment of Arthritis Visual Analogue Scale (PtGA VAS) | Week 24
  The patient's global assessment of disease activity will be measured using 100-mm VAS scale with anchor statements on the left (very well) and on the right (very poorly).
Spondyloarthritis Research Consortium of Canada Enthesitis Index (SPARCC) | Week 24
  The SPARCC Enthesitis Index is a composite score that quantifies the extent of tenderness at 16 sites on a dichotomous basis.
Leeds Enthesitis Index (LEI) | Week 24
  The LEI is an enthesitis index that involves evaluation of tenderness at 6 examination points/sites bilaterally. The LEI score can range between 0 and 6, with higher scores indicating more enthesis sites.
Dactylitis Count | Week 24
  Dactylitis is characterized by diffuse swelling of a finger and/or toe.
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | Weeks 12 and 24
  The BASDAI is a self-administered instrument that measures severity of fatigue/tiredness, spinal and peripheral joint pain, localized tenderness, and morning stiffness. The BASDAI score can range between 0 and 10, with higher scores indicating worse disease control.
Health Assessment Questionnaire-Disability Index (HAQ-DI) | Weeks 12 and 24
  The HAQ-DI is a patient questionnaire that evaluates the degree of disability and pain index over the past week. The HAQ-DI score can range between 0 and 3, with higher scores indicating more disability and pain.
Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) | Weeks 12 and 24
  The FACIT-F is a 13-item measure, which be used to assess fatigue and its impact on daily activities and function in the past 7 days. The FACIT-F score can range between 0 and 52, with higher scores indicating less fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, Principal Investigator — Innovaderm Research Inc.

IPD SHARING:
Plan to Share IPD: No